CLINICAL TRIAL: NCT01651364
Title: A Pilot Study of Cabergoline for the Treatment of Cocaine Dependence
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Thomas Newton, Professor, Baylor College of Medicine
Allocation: Randomized | Model: Parallel | Masking: Quadruple
Other Study IDs: H-27036; DPMC (Other: NIDA); 2630090202 (Other Grant/Funding Number: Baylor Cost Center)
Record Dates: First submitted 2012-02-20; First posted 2012-07-27 (Estimated); Last update posted 2012-07-27 (Estimated); Status verified 2012-07

CONDITIONS: Cocaine Dependence; Cocaine Abuse; Cocaine Addiction; Substance Abuse
Keywords: Cocaine; Cabergoline
MeSH Terms: conditions — Cocaine-Related Disorders; Substance-Related Disorders | interventions — Sugars; Cabergoline

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- Cabergoline (Active Comparator)
  Interventions: Drug: Cabergoline

INTERVENTIONS:
Drug: Placebo — Enrolled volunteers will be randomized on Day 8 to receive placebo (n=2) or study medication (n=8). Placebo serves only to maintain the blind and is not a comparator.
  Other Names: Sugar pill
  Arms: Placebo
Drug: Cabergoline — Enrolled volunteers that receive study medication (n=8) will receive cabergoline 0.25 mg twice weekly.
  Other Names: Dostinex; Cabaser
  Arms: Cabergoline

SUMMARY:
The purpose of this study is to determine the effects of treatment with cabergoline, compared to treatment with placebo, on cocaine induced craving and subjective effects in cocaine-dependent human volunteers.

DETAILED DESCRIPTION:
Secondary aims are to clarify the genetics of substance abuse, potentially leading to improved methods to diagnosis those at risk and to help develop better therapeutic interventions and to develop a new saliva-based test for the detection and measurement of drugs of abuse. As an additional aim, we will also collect blood samples for analyzing a number of genetic polymorphisms.

ELIGIBILITY:
Inclusion Criteria:

* Be English-speaking volunteers who are not seeking treatment at the time of the study.
* Be between 18-55 years of age.
* Meet DSM-IV TR criteria for cocaine dependence; participants may or may not meet criteria for nicotine dependence. Nicotine dependence is allowed but not required because most cocaine users smoke cigarettes.
* Have a self-reported history of using cocaine by the smoked or IV route.
* Have vital signs as follows: supine blood pressure > 100/65 mm Hg. To ensure that subjects will not be at risk from cocaine, the resting pulse must be < 90 bpm and the blood pressure must be < 150 mmHg systolic and < 90 mmHg diastolic.
* Have hematology and chemistry laboratory tests that are within normal (+/- 10%) limits with the following exceptions: a) liver function tests (total bilirubin, ALT, AST, and alkaline phosphatase) ≤ 3 x the upper limit of normal, and b) kidney function tests (creatinine and BUN) within normal limits.
* Have a baseline EKG that demonstrates clinically normal sinus rhythm, clinically normal conduction, and no clinically significant arrhythmias.
* Have a medical history and brief physical examination demonstrating no clinically significant contraindications for study participation, in the judgment of the admitting physician and the principal investigator.
* Females must have a negative urine pregnancy test during screening and at followup, on day 22.
* Provide a negative urine test for cocaine metabolite on Day 1.

Exclusion Criteria:

* Meet DSM IV TR criteria for dependence on drugs other than cocaine or nicotine.
* Have any history or evidence suggestive of seizure disorder or brain injury.
* Have any previous medically adverse reaction to cocaine, including loss of consciousness, chest pain, or epileptic seizure.
* Have a history of heart valve disease.
* Have any evidence from physical exam of heart murmur.
* Have neurological or psychiatric disorders, such as: psychosis, bipolar illness or major depression as assessed by MINI; organic brain disease or dementia assessed by clinical interview; history of any psychiatric disorder which would require ongoing treatment or which would make study compliance difficult; history of suicide attempts within the past year and/or current suicidal ideation/plan.
* Have evidence of clinically significant heart disease or hypertension, as determined by the PI.
* Have evidence of untreated or unstable medical illness including: neuroendocrine, autoimmune, renal, hepatic, or active infectious disease.
* Have symptomatic HIV or are taking antiretroviral medication.
* Be pregnant or nursing. Other females must either be unable to conceive (i.e., surgically sterilized, sterile, or post-menopausal) or be using a reliable form of contraception (e.g., abstinence, birth control pills, intrauterine device, condoms, or spermicide). All females must provide negative pregnancy urine tests before study entry, upon hospital admission, and at the end of study participation.
* Have asthma or currently use theophylline or other sympathomimetics.
* Have any other illness, condition, or use of psychotropic medications, which in the opinion of the PI and/or the admitting physician would preclude safe and/or successful completion of the study.

Criteria for Discontinuation Following Initiation:

* Inability to comply with study procedures.
* Meet discontinuation criteria due to exaggerated response to cocaine, described below.
* Use cocaine prior to randomization.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 11 (Actual)
Dates: Start 2011-07; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
The effects of treatment with cabergoline and cocaine on cardiovascular measures
  Before and after each cocaine infusion, physiologic responses will be closely monitored using repeated HR, BP, and ECG readings. To evaluate safety, a DSMB will meet annually and following any serious AE to examine data as well as any new published information on cabergoline relevant to the project. The number of AEs (including arrhythmias and ECG changes), changes in BP and HR, and changes in mood and psychiatric symptoms (using the BSI, BDI, POMS, and BPRS) will also be assessed throughout the study.

SECONDARY OUTCOMES:
The effects of treatment with cabergoline and cocaine on cocaine-induced craving and subjective effects
  The ability of cabergoline, as compared to placebo, to reduce cocaine-induced craving and to reduce reinforcing effects produced by cocaine will be measured by: 1. VAS, Adjective Scales, and MCQ; 2. Choices for cocaine vs. money in the self-administration assay.

CONTACTS AND LOCATIONS:
Locations (1):
- Michael E. DeBakey VA Medical Center, Houston, Texas, United States